CLINICAL TRIAL: NCT00727467
Title: A Randomised Controlled Trial Evaluating the Effect of an Individual Auditory Cueing Device on Freezing and Gait Speed in People With Parkinson's Disease
Brief Title: A Randomised Controlled Trial (RCT) to Evaluate Use of an Individual Auditory Cueing Device's (IACD's) on Freezing and Gait in People With Parkinson's Disease (PD)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Dr. Emma Stokes, University of Dublin, Trinity College
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5-6-08
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-08

CONDITIONS: Parkinson's Disease
Keywords: auditory cueing device; Parkinson's disease; freezing; gait; mobility
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): On Days 1-8 of the trial, participants in Group A will be given the iPod with some music on the device to allow all participants to become familiar with the device i.e. turning device on and off, increasing and decreasing the volume. They will be instructed to use the device only when sitting at home, and that the device should not be turned on when walking or performing any mobility related or daily tasks.
  On Days 8-15, participants in Group A will be allocated to the 'intervention' phase. Each participant will be given an iPod containing an auditory cue in the form of a continuous metronome beat, individualised to the patient's walking frequency (less 10%).Participants will be instructed to listen to the cueing when they are performing any mobility related tasks. On Days 15-23, participants in Group A will be allocated to the 'control' phase. During this time period, participants will be provided with the iPod shuffle containing no music or metronome beat.
  Interventions: Device: Auditory Cueing Device
- B (Active Comparator): On Days 1-8 of the trial, participants in Group B will be given the iPod with some music on the device to allow all participants to become familiar with the device. They will be instructed to use the device only when sitting at home, and that the device should not be turned on when walking or performing any mobility related or daily tasks.
  On Days 8-15, participants in Group B will be allocated to the 'control' phase. During this time period, participants will be provided with the iPod shuffle containing no music or metronome beat. On Days 15-23, participants in Group B will be allocated to the 'intervention phase'. Each participant will be given an iPod containing an auditory cue in the form of a continuous metronome beat, individualised to the patient's walking frequency (less 10%).Participants will be instructed to listen to the cueing when they are performing any mobility related tasks.
  Interventions: Device: Auditory Cueing Device

INTERVENTIONS:
Device: Auditory Cueing Device — Each participant will be given an iPod containing an auditory cue in the form of a continuous metronome beat, individualised to the patient's walking frequency (less 10%).Participants will be instructed to listen to the cueing when they are performing any mobility related tasks.
  Other Names: iPod shuffle

SUMMARY:
The primary aim of the study is to evaluate the effect of an IACD i.e. Apple iPod-shuffle, on freezing and gait speed in people with a diagnosis of PD through the implementation of a randomised controlled trial. A secondary aim of the study is to evaluate the impact of such a device on the quality of life of people with stroke through the administration of a self-report questionnaire. The IACD will be pre-loaded with an individualised auditory cueing frequency (metronome sound) matched to the walking speed of the individual with PD.

DETAILED DESCRIPTION:
The investigators calculated and pre-loaded 100 baseline frequencies (less 10%) in the sound of a metronome beat in an MP3 format (30 - 130 BPM) [38] onto a DVD-Rom. A user manual was created with a set of instructions that gives each physiotherapist a step-by-step guide on how to calculate the correct beat for their participants and how to successfully upload this beat onto the iPod. In addition physiotherapists in participating centres attended a training session on how to complete the tasks. A pack including the DVD-Rom, user manual, information leaflet and consent was sent to participating centres. Recruitment is due to commence in September 2008.

ELIGIBILITY:
Inclusion Criteria:

* PD
* medically stable
* willing to give informed consent
* freeze at least once per week (minimum score of 2 on item 3 of the FOGQ) for at least 2 seconds(minimum score of 1 on item 4 of FOGQ)
* MMSE Score greater than 24

Exclusion Criteria:

* attending physiotherapy at time of recruitment
* unwilling to give informed consent
* not medically stable
* cognitive impairment (MMSE score less than 24)
* acure co-morbidity that prevents mobility

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-12 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Freezing of Gait Questionnaire | Day 8, Day 15, Day 23 and 3 month follow up

SECONDARY OUTCOMES:
Timed Up and Go Test | Day 8, Day 15, Day 23 and three month follow-up
Modified Falls Efficacy Scale | Day 8, Day 15, Day 23 and three month follow-up
10 Metre Walk Test | Day 8, Day 15, Day 23 and three month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Emma K Stokes, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (3):
- Ireland (3):
  - Cork University Hospital, Cork
  - Royal Hospital Donnybrook, Dublin
  - Saint James's Hospital, Dublin

REFERENCES:
- [Derived] Ledger S, Galvin R, Lynch D, Stokes EK. A randomised controlled trial evaluating the effect of an individual auditory cueing device on freezing and gait speed in people with Parkinson's disease. BMC Neurol. 2008 Dec 11;8:46. doi: 10.1186/1471-2377-8-46. PMID 19077238